CLINICAL TRIAL: NCT06575244
Title: The Effects of a Nurse-led Community-based Sailing Programme on Resilience of School-aged Children With Autism: A Pilot Randomised Controlled Study
Brief Title: The Effects of a Nurse-led Community-based Sailing Programme on Resilience of School-aged Children With Autism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Sailability Hong Kong (Unknown)
Responsible Party: Principal Investigator, Myrian Sze Nga Fan, PhD Candidate, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NTEC-2025-237-T
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Autistic Disorders Spectrum; Child Development
Keywords: Autism spectrum disorder; Children; Sailing; Resilience; Nature-based intervention
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The intervention is guided by the Synergy Model of Resilience, integrating Kolb's theory of experiential learning.
Who Masked: Outcomes Assessor
Masking Description: Due to the limited resources available, the study team has decided to adopt a volunteer-based approach for the blinded outcome assessor. Individuals with relevant experience working with children with autism spectrum disorder (ASD) will be recruited and trained to perform the data collection for the study.
  The researchers recognize the importance of ensuring the reliability and validity of the study's findings. To address this, the volunteer assessors will undergo appropriate training and supervision to equip them with the necessary skills and knowledge to conduct the assessments in a rigorous and unbiased manner.
  By leveraging the expertise and commitment of volunteers with prior experience in the ASD population, the study team aims to overcome the challenge of limited resources and implement the blinded assessment protocol as intended. This approach will help maintain the integrity of the study's methodology and the credibility of the final results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Eligible participants will participate in the nurse-led CBS programme, utilising dinghies with a universal design known for their exceptional stability to prioritize safety. The concrete experience will be introduced through sailing activities. The instructor-to-participant ratio will be 1:6 with a safety boat present. The programme will conclude with participants receiving a certificate of participation.
  Interventions: Other: Community-based sailing
- Controlled group (Placebo Comparator): Participants in the attention control group will participate in crafting activities. These activities will match the time and attention dedicated by the intervention group but are designed to have no impact on resilience.
  Interventions: Other: Crafting activities

INTERVENTIONS:
Other: Community-based sailing — A nurse-led community-based sailing programme is validated by an expert panel including professionals from various fields, such as a registered nurse, academia, and qualified sailing instructors, delivered in a group of 6 participants, incorporating experiential learning, with the aid of materials including dinghies with Universal design, safety boats, buoys, buoyancy aids, supplementing with a waterproof sailing booklet. The intervention is developed and facilitated by a registered nurse (principal investigator).
  Arms: Intervention group
Other: Crafting activities — Participants in the attention control group will participate in crafting activities. Activities match the time and attention dedicated by the intervention group. Activities are designed to have no impact on resilience.
  Arms: Controlled group

SUMMARY:
The goal of this pilot RCT is to evaluate the feasibility and acceptability of the community-based sailing program and to assess the preliminary effects before the main RCT, given the literature on sailing for children with ASD has not yet been established.

Does intervention improve the resilience of participants? Does intervention improve the quality of life, self-esteem, depressive symptoms, and social functioning outcomes of participants?

Researchers will compare the effect of community-based sailing to the attention control group at baseline, following randomisation, and post-intervention

Participants will:

Participants in the intervention group will participate in a nurse-led community-based sailing programme over six days, with each day consisting of 4 sessions, each lasting an hour, for a total of 24 hours.

Participants in the attention control group will engage in crafting activities with minimal difficulty, focusing on maintaining attention without any emotional or reflective discussions.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental condition that typically emerges in early childhood, characterized by persistent deficits in social communication and interaction, with the presence of restricted, repetitive patterns of behaviour, interests, or activities. This study seeks to address the outcome gap in the literature, the resilience of children with ASD, and expand their natural environment to include nature and the community through nature-based interventions (NBIs).

Considering the limited generalizability of autism research findings among children due to the expanded definition of the autism spectrum in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), which merged previous diagnostic labels into one spectrum, translating knowledge into practice becomes challenging. Therefore, a stratification approach is adopted to examine the resilience (Primary outcomes), along with secondary outcomes, including QoL, depressive symptoms, self-esteem, and social functioning based on synthesis from prior studies. A study conducted revealed that school-aged children with ASD in inclusive education significantly exhibited more depressive symptoms, lower QoL, lower resilience, and lower self-esteem. Where resilience is identified as a significant mediator in the association between depressive symptoms and psychosocial health, highlighting the potential of resilience-focused interventions in enhancing resilience and supporting mental health.

Existing community-based sailing (CBS) programs, led by qualified sailing instructors and provided to individuals regardless of ability to foster social connection and overall well-being in the community, hold potential as promising nature-based, resilience-focused recreational activities that incorporate experiential learning. A qualitative study highlighted the positive experience among school-aged children with ASD in inclusive education, where resilience emerged to be a key aspect. This study highlights a critical gap in that many children do not understand resilience and perceive their sailing experience merely as recreational. Thereafter, the proposed study aims to develop and evaluate a nurse-led CBS program to enhance their resilience by recognising the nursing expertise in interprofessional collaboration within a community-based approach.

The proposed study follows the Medical Research Council (MRC)/ National Institute for Health and Care Research (NIHR) framework for developing and evaluating complex interventions. This study will employ a randomized controlled trial (RCT) with an assessor-blind design, in collaboration with the community-based charity organization Sailability Hong Kong, recruiting 36 children with autism aged 7 to 12 years. The results will be analyzed using the Generalized Estimating Equation (GEE) model, following the intention-to-treat (ITT) principle to ensure the reliability of findings.

This pilot study aims to assess the feasibility and acceptability and to evaluate the initial effects of the nurse-led CBS programme on the resilience of school-aged children with ASD.

The study hypothesizes that in comparison to the control group with attention controlled group, school-aged children with ASD in inclusive education who participate in the intervention group will exhibit (1) increased levels of resilience, (2) improved QoL, (3) reduced depressive symptoms, (4) enhanced self-esteem, (5) improved social functioning immediately after the intervention.

The innovative aspect of this study lies in utilizing CBS as a therapeutic approach aimed at enhancing the resilience of children with ASD in supporting their mental health. This research is original and innovative, building on previous evidence, including systematic reviews, cross-sectional studies, qualitative studies, and conceptual model development. It seeks to bridge the research gap in resilience.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 7 and 12,
2. have a confirmed diagnosis of ASD,
3. be enrolled in inclusive education school,
4. possess the ability to complete the questionnaire in Chinese,
5. be able to communicate in Chinese.

Exclusion Criteria:

* With sailing experience,
* With a history of severe motion sickness symptoms.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Resilience | Pre-intervention, Post-intervention (within 1 week immediately after intervention)
  The Resilience Scale-14 (RS-14) consists of 14 items assessing personal competence, acceptance of self, and life. Each item is rated on a 7-point Likert scale, ranging from "strongly disagree" to "strongly agree." The total possible scores on the RS-14 range from 14 to 98, with higher scores indicating higher levels of resilience. The Chinese version of the RS-14 has been validated for evaluating the resilience of young adolescents in Hong Kong. It demonstrates good internal consistency, with a Cronbach's alpha coefficient of 0.86.

SECONDARY OUTCOMES:
Depressive symptoms | Pre-intervention, Post-intervention (within 1 week immediately after intervention)
  The Chinese version of the Center for Epidemiologic Studies Depression Scale for Children (CES_DC) comprises 20 standardized items designed to assess depressive symptoms in children across three domains: emotional, cognitive, and behavioral-related components of depression. Participants rate the frequency of each symptom experienced during the previous week on a 4-point Likert scale. Scores range from 0 to 3 (0 = not at all, 1 = a little, 2 = some, and 3 = a lot) for each item. The total possible CES-DC scores range from 0 to 60, with higher scores indicating a greater number of symptoms. A score of 16 or higher suggests the presence of depressive symptoms. The Chinese version of the CES-DC has been validated for use in children in Hong Kong and exhibits adequate internal consistency, as indicated by a Cronbach's alpha coefficient above 0.8.
Self-esteem | Pre-intervention, Post-intervention (within 1 week immediately after intervention)
  Rosenberg's Self-Esteem Scale (RSES) is a widely used tool for measuring global self-worth in both positive and negative aspects of self-perception. The scale consists of 10 items and has been employed with children. Participants responded to the items using a 4-point Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). Total scores on the RSES range from 10 to 40, with higher scores indicating higher levels of self-esteem. The Chinese version of the RSES has demonstrated internal consistency, with a Cronbach's alpha coefficient of 0.78 in a study conducted in Hong Kong.
QoL | Pre-intervention, Post-intervention (within 1 week immediately after intervention)
  The Pediatric Quality-of-Life Inventory 4.0 Generic Core Scale (PedsQL™) is utilized to assess participants' perception of their quality of life (QoL) across various domains, including the impact of disease and treatment on physical functioning (eight items), emotional functioning (five items), social functioning (five items), and school functioning (five items). Participants rate the extent to which each item has been problematic over the past month, using a scoring system ranging from 0 to 4 (0 = never, 1 = almost never, 2 = sometimes, 3 = often, and 4 = almost always). The items are then reverse scored and linearly transformed to a 0-100-point scale, with higher scores indicating better health-related QoL. The Chinese version of the PedsQL™ comprises 23 items and has been validated, demonstrating a Cronbach's alpha coefficient of 0.90.
Social functioning outcomes | Pre-intervention, Post-intervention (within 1 week immediately after intervention)
  The 2nd edition of the Social Responsiveness Scale (SRS-2) is a questionnaire, consisting of 65 items that measure the severity of symptoms associated with ASD. Participants' parents rate them on a 4-point Likert scale ranging from 0 (never true) to 3 (almost always true). The SRS includes five subscales: social awareness, social cognition, social communication, social motivation, and autistic mannerisms. These subscales help assess different aspects of social functioning. The questionnaire also provides a total score, with higher scores indicating higher levels of impairment. The SRS demonstrates strong internal consistency, with a Cronbach's alpha coefficient of .97. The Chinese version of the RSES has demonstrated internal consistency, with a Cronbach's alpha coefficient of 0.9 in a study conducted in China.

CONTACTS AND LOCATIONS:
Overall Officials: Myrian Sze Nga Fan, MSc, Principal Investigator — Chinese University of Hong Kong; Professor William Ho Cheung Li, PhD, Study Chair — Chinese University of Hong Kong; Professor Laurie Long Kwan Ho, PhD, Study Director — Chinese University of Hong Kong; Chair Sek Ying Professor Chair Sek Ying, PhD, Study Chair — Chinese University of Hong Kong
Locations (1):
- The Nethersole School of Nursing, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The research team does not have plans to proactively or automatically make the individual participant data (IPD) from this study available to other researchers. However, the IPD may be shared upon request, provided that the requesting party has a valid scientific or medical rationale and obtains the necessary approval from the research team.
  Any requests for access to the study's IPD will be reviewed on a case-by-case basis by the research team. Factors that will be considered in evaluating such requests include:
  * Scientific merit and validity of the proposed use of the data
  * Qualifications and track record of the requesting researcher or research team
  * Alignment with the original study objectives and participants' consent